CLINICAL TRIAL: NCT01360944
Title: An Investigator-blind, Controlled Exploratory Study to Assess the Efficacy and Safety of Different Concentrations of Active Ingredients in the Project LAS 41004 Compared to a Bland Ointment and to Active Control in a Psoriasis- Plaque- Test
Brief Title: Exploratory Study to Investigate Efficacy of LAS41004 in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Almirall, S.A. (Industry)
Collaborators: Sciderm GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H553000-1006; 2011-000186-13 (EudraCT Number)
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Psoriasis
Keywords: PPT, topical, psoriasis
MeSH Terms: conditions — Psoriasis; Ceroid lipofuscinosis, neuronal 1, infantile

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- LAS 41004, variant 1, once daily (Experimental): variant 1, once daily
  Interventions: Drug: LAS41004
- LAS41004, variant 2, once daily (Experimental): variant 2, once daily
  Interventions: Drug: LAS41004
- LAS41004, variant 3, once daily (Experimental): variant 3, once daily
  Interventions: Drug: LAS41004
- LAS41004, variant 4, once daily (Experimental): variant 4, once daily
  Interventions: Drug: LAS41004
- LAS41004, variant 5, once daily (Experimental): variant 5, once daily
  Interventions: Drug: LAS41004
- LAS41004, variant 6, once daily (Experimental): variant 6, once daily
  Interventions: Drug: LAS41004
- reference (Placebo Comparator): once daily, 100microgram
  Interventions: Drug: reference
- reference, once daily (Active Comparator): once daily
  Interventions: Drug: reference

INTERVENTIONS:
Drug: LAS41004 — once daily, topical, 100 microgram
  Arms: LAS 41004, variant 1, once daily; LAS41004, variant 2, once daily; LAS41004, variant 3, once daily; LAS41004, variant 4, once daily; LAS41004, variant 5, once daily; LAS41004, variant 6, once daily
Drug: reference — once daily, 100 microgram
  Arms: reference; reference, once daily

SUMMARY:
The aim of the exploratory study is to compare the dose-related efficacy of LAS41004 in a Psoriasis Plaque Test (PPT).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients between 18 and 75 years of age with a diagnosis of stable plaque-type psoriasis (psoriasis vulgaris) for at least 12 months
* Psoriatic plaques that are suitable to be defined as target area lesions by the following criteria:

oPsoriatic plaques must be located on the trunk and/or extremities. Plaques that are located on the head (incl. scalp), palms, sole of the feet, intertriginous or genitoanal areas are not suitable as target areas

* Comparable psoriatic plaques with at least "2" in each score (range 0-4) for the three distinct signs: scaling, erythema and induration
* No more than 3 points difference in total score (= sum of scores for scaling, erythema and induration; Range 0-12) of the chosen comparable psoriatic plaques
* Enough surface area to the psoriatic plaque to define eight clearly distinguishable (minimum distance between test areas: 1cm) test areas of at least 1 cm² size - Effective contraceptive methods for the duration of the study and for the 4 weeks after study drug discontinuation, for a patient of childbearing potential.

Key Exclusion Criteria:

* Too small a body surface area covered with psoriasis plaques that meet the specified inclusion criteria
* Any condition that may interfere with the study assessments or ultrasound measurements of the skin and/or may have an influence on the skin immune response (incl. open wounds)
* Current diagnosis of guttate, erythrodermic or pustular psoriasis
* Patients who have received any topical anti-psoriatic drug in the test area within the last 2 weeks before treatment with the IMP.
* Patients who have received topical products in the test area containing DEET (N,N-diethyl-m-polyamide), a common component of insect repellent products within 1 week before treatment with the IMP.
* Patients who have received systemic biologics within the last 6 months before treatment with the IMP or any systemic antipsoriatic treatment (corticosteroids, ciclosporin, methotrexate, fumaric acid esters, acitretin etc)within the last 3 months before treatment with the IMP.
* Significant skin diseases other than plaque-type psoriasis (psoriasis vulgaris), including but not limited to: skin disease due to tuberculosis or syphilis, rosacea, perioral dermatitis, acne vulgaris, skin atrophy, striae distensae, increased fragility of skin blood vessels, ichthyosis, ulcers, wounds and reaction after vaccination
* Significant skin infections (including but not limited to: herpes, varicella, mycotic skin infections, bacterial skin infections or parasitic skin infections)
* Excessive sunlight exposure within 28 days prior to study entry and during the conduct of the study
* Usage of any topical formulation (incl. cosmetics, emollients, etc) on the designated target areas during the course of the study
* Vitamin A intake > 15,000 IU/day

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Decrease in thickness of infiltration | Day 1 (baseline) vs day 15 day (final)
  measurement will be performed by ultrasound, comparing data from baseline (day1) vs end of trial (day15)

SECONDARY OUTCOMES:
Change in clinical score | day 1 (baseline) vs day 15 (final)
  scoring of total symptom score (0 - 12)will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Change in erythema score | day1 (baseline) vs day 15 (final)
  scoring of erythema (0-4) will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Change in Induration score | day 1 (baseline) vs day 15 (final)
  scoring of induration (0-4) will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)
Change in Scaling score | day 1 (baseline) vs day 15 (final)
  scoring of scaling (0-4) will be performed by investigator, comparing data from baseline (day1) vs end of trial (day15)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Willers, MD, Study Director — Almirall Hermal
Locations (1):
- Investigational site, Mahlow, Germany